CLINICAL TRIAL: NCT01450202
Title: Carbon Dioxide Insufflation During Colonoscopy With Consecutive EGD is Safe and Decreases Abdominal Pain in Sedated Outpatients: a Randomized, Double-blind, Controlled Trial
Brief Title: Safety and Efficacy of Carbon Dioxide Insufflation During Colonoscopy With Consecutive Esophagogastroduodenoscopy in Reduction of Abdominal Pain in Sedated Outpatients
Acronym: COCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Eun Hee Seo, MD, principal investigator, Inje University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Oct 2011-01
Record Dates: First submitted 2011-10-04; First posted 2011-10-12 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Pain
Keywords: Carbon dioxide insufflation; Colonoscopy; Esophagogastroduodenoscopy; Bowel insufflation; Postprocedure pain; Pain Due to Certain Specified Procedures
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air insufflation, colonoscopy, esophagogastroduodenoscopy (Placebo Comparator)
  Interventions: Other: bowel insufflation gas
- CO2 insufflation, colonoscopy, esophagogastroduodenoscopy (Active Comparator)
  Interventions: Other: bowel insufflation gas

INTERVENTIONS:
Other: bowel insufflation gas — air insufflation, during colonoscopy and esophagogastroduodenoscopy
  Arms: Air insufflation, colonoscopy, esophagogastroduodenoscopy
Other: bowel insufflation gas — CO2 insufflation, during colonoscopy and esophagogastroduodenoscopy
  Arms: CO2 insufflation, colonoscopy, esophagogastroduodenoscopy

SUMMARY:
Compared with performing each procedure individually, performing two combined procedures such as colonoscopy consecutive Esophagogastroduodenoscopy (EGD) cause more bowel gases, abdominal distension and post-procedure pain because of longer procedure time related to more bowel insufflated gas than one procedure. To the best of the investigators knowledge, there has been no randomized controlled trial of CO2 versus air for insufflations during combined two procedures, colonoscopy with consecutive EGD. And there are a few well randomized trials concerned CO2 insufflation in patients receiving sedation during colonoscopy.

The aim of the present study was to evaluate the efficacy of CO2 in reducing post-procedural abdominal pain and distension during colonoscopy consecutive EGD and to confirm the safety of CO2 insufflation when it is used during procedure in sedated outpatients.

ELIGIBILITY:
Inclusion Criteria:

* outpatients between the ages of 18 and 70 years who are scheduled for colonoscopy with consecutive EGD

Exclusion Criteria:

* age < 18 or > 70 years
* pregnancy
* breast feeding
* chronic obstructive lung disease (COPD)
* known CO2 retention and refusal to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
post-procedural pain | 3 months
  The primary end point of the study was to assess post-procedural pain according to VAS scale

SECONDARY OUTCOMES:
abdominal distention | 3 months
  abdominal distention using measurement of patient waist circumferences
ETCO2 | 3 months
  Measure ETCO2 using nasal cannula

CONTACTS AND LOCATIONS:
Locations (1):
- Haeundae Paik Hospital, Busan, South Korea